CLINICAL TRIAL: NCT02293382
Title: A Retrospective Chart Review of Deceased Patients With Mucopolysaccharidosis Type IIIB
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NGLU-NH01
Record Dates: First submitted 2014-11-03; First posted 2014-11-18 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: MPS IIIB (Sanfilippo Syndrome)
Keywords: MPS IIIB; Mucopolysaccharodosis III; Mucopolysaccharidosis type IIIB; Sanfilippo Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to perform a retrospective chart review to generate data to evaluate the clinical characteristics and course of disease progression of MPS IIIB.

ELIGIBILITY:
Inclusion Criteria:

1. The deceased patient was diagnosed with MPS IIIB as determined by either of the following:

   1. Documented deficiency of NAGLU enzyme activity.
   2. Documented functionally-relevant mutations in both alleles of the NAGLU gene.
2. Patient's parent or legal guardian provides informed consent (unless the requirement for informed consent is waived by local regulations).
3. The availability of pre-defined information in the patient's clinical chart:

Exclusion Criteria:

There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 deceased patients with MPS IIIB
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of disease presentation and the course of disease progression including the end stage of the disease in patients with MPS IIIB, assessed from medical history data obtained by retrospective chart review of deceased patients. | N/A as this is a retrospective chart review of deceased patients
  Data obtained by retrospective chart review will include medical history data including patient demographics, disease manifestation onset, clinical history, diagnostic tests and treatments for MPS IIIB, supportive interventions/medications, clinical chemistry and haematology results, anthropometric data, radiology results, and autopsy findings.

CONTACTS AND LOCATIONS:
Locations (5):
- Pittsburgh, Pennsylvania, United States
- Porte Alegre, Brazil
- Amsterdam, Netherlands
- Barcelona, Spain
- Birmingham, United Kingdom